CLINICAL TRIAL: NCT03511417
Title: Aging and Speech Perception in Complex Listening Environments
Brief Title: The Effectiveness of Over the Counter Hearing Products for Middle-Aged Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the delay in establishing FDA regulations for over-the-counter hearing aids
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Karen Helfer, Professor and Chair, University of Massachusetts, Amherst
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01DC012057-06 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-04-27 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss, Functional
MeSH Terms: conditions — Hearing Loss, Functional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Middle-aged adults (Experimental): Participants will use an over-the-counter hearing device in one ear until asymptotic speech perception performance is noted (maximum 12 weeks). The same individuals will use over-the-counter hearing devices in each ear until asymptotic performance is noted (the order of these two phases will be randomized across participants). They will be asked to use these devices at least 4 hours/day.
  Interventions: Device: over-the-counter hearing device

INTERVENTIONS:
Device: over-the-counter hearing device — Individuals will use commercially-available over-the-counter hearing devices for specified periods of time.

SUMMARY:
The investigators will examine the effectiveness of selected over-the-counter personal sound amplifiers in addressing functional hearing problems in middle-aged listeners with mild hearing loss. Many people are unlikely to pay several thousand dollars for hearing aids but they likely would be more willing to try a possible solution that is less expensive. When faced with counseling these individuals, audiologists are at a loss regarding whether or not to suggest that they try this type of technology, since there is virtually no research available to verify that these devices actually are helpful, particularly for individuals with mild hearing loss. The hypothesis being tested is that personal sound amplifiers can improve functional hearing and decrease cognitive load in complex auditory environments.

DETAILED DESCRIPTION:
The field trials in this project will require you to use OTC hearing devices for a specified period of time in both ears simultaneously, and in just one ear, with periodic lab-based re-evaluation. Each field trial will continue until asymptotic performance is identified (up to a maximum of 12 weeks). You will return to the lab for assessment every 2 weeks. During each visit, speech perception and subjective listening effort will be assessed. Depending upon the specific field trial, the investigators also will complete measures of cognitive load (via dual-task paradigms), spatial release from masking, and localization ability during each lab visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-64 years
* Mild to moderate high frequency hearing loss
* Learned English as a first language

Exclusion Criteria:

* Previous use of hearing aids
* Hearing loss/problems attributed to factors other than aging
* History of: neurologic disorder, middle-ear disease
* Score of < 26 on the Montreal Cognitive Assessment

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Speech Perception | every two weeks until asymptotic performance is noted (up to 12 weeks)
  The change in the ability to understand sentences presented in background noise
Cognitive Load | every two weeks until asymptotic performance is noted (up to 12 weeks)
  The change in the ability to remember speech that has previously been presented in background noise
Localization Ability | every two weeks until asymptotic performance is noted (up to 12 weeks)
  The change in the ability to indicate where a sound is coming from when presented in background noise
Self-Perceived Listening Effort | every two weeks until asymptotic performance is noted (up to 12 weeks)
  Changes in how difficult it is to understand speech in background noise

SECONDARY OUTCOMES:
Self-perceived hearing device benefit | daily during field trial (up to 12 weeks)
  The situations in which participants find the hearing aids to be beneficial
Overall perceived benefit from hearing device | every two weeks until asymptotic performance is noted (up to 12 weeks)
  The extent to which participants believe the hearing devices help them

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No